CLINICAL TRIAL: NCT02184871
Title: Next Generation Sequencing in Intrahepatic Cholangiocarcinoma (ICC) According to the Stratification of the Risk Factors
Brief Title: Next Generation Sequencing in Intrahepatic Cholangiocarcinoma
Acronym: EtherBil
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Giovanni Brandi, Prof, MD, PhD, University of Bologna
Other Study IDs: 21/2014/U/Tess
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; RNAseq; risk factors; asbestos
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue samples will be immediately collected after surgery: one part will be suspended in RNAlater to prevent RNA degradation and stored at -20°C, the other will be formalin-fixed and paraffin-embedded for histopathology examination and evaluation of asbestos fibers. For each patient enrolled, peripheral blood will be also collected and stored at -20°C. Total RNA and genomic DNA will be extracted from tumor tissue and peripheral blood and stored at -80°C until use.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intrahepatic cholangiocarcinoma: Patients committed to surgery and stratified according to exposure to different risk factors for ICC, basing on modified ReNaM questionnaire.
  Interventions: Other: exposure to different risk factors and molecular assessment

INTERVENTIONS:
Other: exposure to different risk factors and molecular assessment

SUMMARY:
The aim of the present study is to perform a comprehensive molecular characterization of intrahepatic cholangiocarcinoma (ICC) in patients exposed to well-known or putative risk factors (such as asbestos) for this malignancy, in order to identify possible "molecular signatures" associated to such different risk factors.

DETAILED DESCRIPTION:
Exposure to distinct risk factors of the enrolled ICC patients will be assessed by modified ReNaM questionnaire. Molecular characterization of ICC tissue samples will be carried out by RNAseq. Briefly, after surgical resection tissue samples will be immediately suspended in RNAlater. RNAseq analysis will be performed on the Illumina HiScanSQ platform. Any possible mutations identified by RNAseq will be validated by Sanger sequencing. Putative identified fusion transcripts will be confirmed by RT-PCR, using specific primers pairs located on the sequences from the exons of the two putative fusion genes. Variations in gene expression will be validated by the real-time PCR. The bioinformatic analysis will be made by using CentOS5 Server. For evaluation of asbestos fibers in tumor tissues, samples embedded in paraffin will be incinerated and then analyzed in a scanning electron microscope and by EDS spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients having a confirmed diagnosis of ICC resected;
* patients who have signed the informed consent;
* patients (males or females) who are at least 18 years old.

Exclusion Criteria:

* patients who have been treated with any medical treatment (chemotherapy or experimental standard) or with radiotherapy during the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICC patients candidate for curative-intent surgery, for a total of 45 subjects. For each patient enrolled, histological examination of tumor tissue specimen will be performed in order to confirm ICC diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Identification of molecular biomarkers in ICC patients exposed to different risk factors. | 3 years
  For each patient enrolled, molecular profile of ICC tissue samples will be correlated to the anamnestic data collected by modified ReNaM questionnaire. For bio-informatic analysis, the collected data will be analyzed in order to identify signals that significantly deviate from the expected SNVs distribution in the general population, then analyzing the presence of clustering for the selected genes group. A two-way unsupervised hierarchical clustering analysis will be run to assess gene expression in the study groups (exposed / unexposed to the different risk factors). Random permutation test will be also conducted to assess the presence of genes whose expression is different in the study groups. Statistical analyses will be conducted using the R software (R Foundation and for Statistical Computing).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Brandi, Principal Investigator — University of Bologna
Locations (1):
- Policlinico S.Orsola- Malpighi, S.S.D. Oncologia Medica- Biasco, Bologna, BO, Italy